CLINICAL TRIAL: NCT00669669
Title: Benzylguanine-Mediated Tumor Sensitization With Chemoprotected Autologous Stem Cells for Patients With Malignant Gliomas
Brief Title: O6-Benzylguanine-Mediated Tumor Sensitization With Chemoprotected Autologous Stem Cell in Treating Patients With Malignant Gliomas
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to loss in funding.
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000.00; NCI-2013-00701 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 8357; 2000.00 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1709046 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2008-04-29; First posted 2008-04-30 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-01

CONDITIONS: Glioblastoma; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Radiotherapy, Conformal; Carmustine; carmustine, poliferprosan 20 drug combination; Filgrastim; Granulocyte Colony-Stimulating Factor; Radiotherapy, Intensity-Modulated; O(6)-benzylguanine; plerixafor; ferric pyrophosphate; Proton Therapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, autologous stem cell transplant) (Experimental): See Detailed Description
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carmustine; Biological: Filgrastim; Procedure: In Vitro-Treated Peripheral Blood Stem Cell Transplantation; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: O6-Benzylguanine; Drug: Plerixafor; Radiation: Proton Beam Radiation Therapy; Drug: Temozolomide

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D conformal IMRT
  Other Names: 3-dimensional radiation therapy; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous in vitro-treated peripheral blood stem cell transplant
  Other Names: Autologous Stem Cell Transplantation
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; Gliadel; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Biological: Filgrastim — Given SC
  Other Names: Filgrastim XM02; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tbo-filgrastim; Tevagrastim
Procedure: In Vitro-Treated Peripheral Blood Stem Cell Transplantation — Undergo autologous in vitro-treated peripheral blood stem cell transplant
  Other Names: in vitro-treated PBPC transplantation; in vitro-treated peripheral blood progenitor cell transplantation
Radiation: Intensity-Modulated Radiation Therapy — Undergo 3D conformal IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: O6-Benzylguanine — Given IV
  Other Names: 6-O-BENZYLGUANINE; O(6)-Benzylguanine
Drug: Plerixafor — Given SC
  Other Names: AMD 3100; JM-3100; Mozobil; SDZ SID 791
Radiation: Proton Beam Radiation Therapy — Undergo proton beam radiation therapy
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac

SUMMARY:
This phase I/II trial studies the side effects and best dose of temozolomide when given together with radiation therapy, carmustine, O6-benzylguanine, and patients' own stem cell (autologous) transplant in treating patients with newly diagnosed glioblastoma multiforme or gliosarcoma. Giving chemotherapy, such as temozolomide, carmustine, and O6-benzylguanine, and radiation therapy before a peripheral stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. Giving colony-stimulating factors, such as filgrastim or plerixafor, and certain chemotherapy drugs, helps stem cells move from the bone marrow to the blood so they can be collected and stored. Chemotherapy or radiation therapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy and radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and feasibility of infusing autologous granulocyte colony-stimulating factor (G-CSF) (filgrastim) mobilized stem cells transduced with a Phoenix-gibbon ape leukemia virus (GALV)-pseudotype vector expressing methylguanine methyltransferase (MGMT) (P140K).

II. Define the dose of BCNU (carmustine) that results in efficient engraftment of gene modified cells when given with peripheral blood stem cell support.

SECONDARY OBJECTIVES:

I. Determine the engraftment of gene-modified cells after conditioning with BCNU.

II. Determine the ability to select gene-modified cells in vivo with this regimen.

III. Evaluate the molecular and clonal composition of gene-modified cells after chemotherapy with temozolomide.

IV. Observe patients for clinical anti-tumor response.

V. Determine the correlation of the level of MGMT (P140K) marking with toxicity, temozolomide dose achieved, and response.

VI. Characterize the toxicity associated with this regimen.

OUTLINE: This is a phase I, dose-escalation study of temozolomide followed by a phase II study.

PART I: Within 35 days of surgery, patients undergo 3 dimensional (3D) conformal intensity-modulated radiation therapy (IMRT) or proton beam radiation therapy daily 5 days per week for 6 weeks. Patients receive filgrastim subcutaneously (SC) on days -7 to -3 and begin stem cell collection on the 4th day of filgrastim administration (up to 3 apheresis). Patients may also receive plerixafor SC on days -5 to -3. The CD34+ stem cells are separated from the patient's stem cells and they are transduced with Phoenix-RD114 pseudotype vector (retrovirus). One day after apheresis is completed, patients receive carmustine intravenously (IV) over 3 hours followed 2 hours later by temozolomide orally (PO). At least twenty-four hours after completion of carmustine and temozolomide, patients undergo reinfusion of genetically-modified stem cells.

PART II: Beginning approximately 4 weeks after completion of Phase 1 of the study, patients receive O6-benzylguanine IV continuously over 48 hours followed by temozolomide PO within 1 hour. Treatment may repeat at least every 28 days for a total of 24 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 1-3 months for 2 years, every 3-6 months for 3 years, and then annually thereafter for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glioblastoma multiforme or gliosarcoma
* The patient or legal guardian must be able to comprehend the informed consent form and sign prior to patient enrollment
* Karnofsky performance status at time of study entry must be >= 70%
* Life expectancy of >= 3 months
* Patients must agree to undergo repeat clinical neurological examinations and brain magnetic resonance imaging (MRI) with appropriate contrast after every other cycle of chemotherapy
* White blood cell (WBC) > 3000/ul
* Absolute neutrophil count (ANC) > 1500/ul
* Platelets > 100,000/ul
* Hemoglobin > 10 gm/100ml
* Total and direct bilirubin < 1.5 times upper limit of laboratory normal
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) =< 3 times upper limit of laboratory normal
* Alkaline phosphatase =< 3 times upper limit of laboratory normal
* Blood urea nitrogen (BUN) < 1.5 times upper limit of laboratory normal
* Serum creatinine < 1.5 times upper limit of laboratory normal
* Left ventricular ejection fraction (LVEF) >= 40%, however, subjects with a LVEF in the range of 40-49% should have cardiology clearance prior to intervention
* MGMT promoter methylation analysis of surgically resected tumor or tumor biopsy must demonstrate an unmethylated or hypomethylated MGMT promoter status

Exclusion Criteria:

* Patients with cardiac insufficiency and a LVEF of < 40%; history of coronary artery disease or arrhythmia, which has required or requires ongoing treatment
* Patients with active pulmonary infection and/or pulse oximetry < 90% and a corrected diffusion capacity of the lung for carbon monoxide (DLCO) < 70% of predicted
* Active systemic infection
* Patients who are human immunodeficiency virus (HIV) positive
* Pregnant or lactating women; a beta-human chorionic gonadotropin (HCG) level will be obtained from women of childbearing potential; fertile men and women should use effective contraception
* Previous chemotherapy for any malignancy including temozolomide, dacarbazine (DTIC) or prior nitrosourea
* Diabetes mellitus
* Bleeding disorder
* Methylated or hypermethylated MGMT promoter status within tumor tissue
* Medical or psychiatric condition which in the opinion of the protocol chairman would compromise the patient's ability to tolerate this protocol
* Prior interstitial radiotherapy, stereotactic or gamma knife surgery or implanted BCNU-wafers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-02-25 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Kiem, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Adair JE, Johnston SK, Mrugala MM, Beard BC, Guyman LA, Baldock AL, Bridge CA, Hawkins-Daarud A, Gori JL, Born DE, Gonzalez-Cuyar LF, Silbergeld DL, Rockne RC, Storer BE, Rockhill JK, Swanson KR, Kiem HP. Gene therapy enhances chemotherapy tolerance and efficacy in glioblastoma patients. J Clin Invest. 2014 Sep;124(9):4082-92. doi: 10.1172/JCI76739. Epub 2014 Aug 8. PMID 25105369

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Autologous Stem Cell Transplant)
Started | 12
Completed | 11
Not Completed | 1
Not completed — To late to start treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, Autologous Stem Cell Transplant)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Dose-limiting Toxicity (DLT)
Description: Defined as any grade 4 nonhematopoietic toxicity that is likely related to the investigational procedures (Part I)
Time Frame: Up to 6 weeks after infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Autologous Stem Cell Transplant)
Number analyzed (Participants) | 11
Participants | 1

2. Primary Outcome: Number of Participants With Retrovirus or Leukemia
Description: Replication competent retrovirus or diagnosis of leukemia
Time Frame: Up to 2 years after infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Autologous Stem Cell Transplant)
Number analyzed (Participants) | 11
Participants | 0

3. Secondary Outcome: Response Rate
Description: Number of patients with reduction in tumor burden of a predefined amount
Time Frame: Up to 66 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Autologous Stem Cell Transplant)
Number analyzed (Participants) | 11
Participants | 1

4. Secondary Outcome: Duration of Response
Description: From the onset of temozolomide to the date at which unequivocal disease progression, assessed up to 65 months.
Time Frame: Up to 65 months
Population: Reduction in number of patients assessed relative to total patients enrolled is due to some patient's disease progressing prior to start of temozolomide.
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Chemotherapy, Autologous Stem Cell Transplant)
Number analyzed (Participants) | 6
months | 4.5 [2.5 to 65.2]

5. Secondary Outcome: Time to Progression
Description: From the first day of treatment (transplant) until unequivocal progression is documented, assessed up to 66 months.
Time Frame: Up to 66 months.
Population: as for outcome 4
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Chemotherapy, Autologous Stem Cell Transplant)
Number analyzed (Participants) | 6
months | 5.5 [3.8 to 66.1]

6. Secondary Outcome: Number of Participants That Survived
Description: From the first day of treatment until death, assessed up to 74 months.
Time Frame: Up to 74 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Autologous Stem Cell Transplant)
Number analyzed (Participants) | 11
Participants | 0

7. Secondary Outcome: Number of Participants With Chemoprotection
Description: assessed by the ability to increase the Temozolomide dose beyond 472 mg/m^2
Time Frame: Up to 66 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Autologous Stem Cell Transplant)
Number analyzed (Participants) | 11
Participants | 2

8. Secondary Outcome: Number of Participants With Chemoselection
Description: assessed by the increase in peripheral blood Vector Copy Number (VCN), the average copies of integrated transgene per cell, after chemotherapy
Time Frame: Up to 59 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Autologous Stem Cell Transplant)
Number analyzed (Participants) | 11
Participants | 4

9. Secondary Outcome: Gene Transfer Efficiency
Description: Assessed by gene marking in peripheral blood prior to chemoselection. Gene marking is assessed in whole blood by quantitative PCR and reported as a vector copy number (VCN) or the average copies of integrated transgene per cell. The units here will be reported as copies/cell.
Time Frame: Up to 59 months
Measure: Mean (Standard Error); unit: copies/cell
Arm/Group | Treatment (Chemotherapy, Autologous Stem Cell Transplant)
Number analyzed (Participants) | 11
copies/cell | 0.78 (0.11)

10. Secondary Outcome: Gene Transfer Efficiency After Chemotherapy
Description: Assessed by gene marking in peripheral blood after chemoselection. Gene marking is assessed in whole blood by quantitative PCR and reported as a vector copy number (VCN) or the average copies of integrated transgene per cell. The units here will be reported as copies/cell.
Time Frame: Up to 59 months
Measure: Mean (Standard Error); unit: copies/cell
Arm/Group | Treatment (Chemotherapy, Autologous Stem Cell Transplant)
Number analyzed (Participants) | 11
copies/cell | 0.50 (0.13)

ADVERSE EVENTS:
Time Frame: Serious and other Adverse Events are collected through study completion, on average 2 years. All cause mortality was assessed up to 7 years.
Arm/Group | Treatment (Chemotherapy, Autologous Stem Cell Transplant)
All-Cause Mortality (participants affected / at risk) | 11/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Autologous Stem Cell Transplant) (N=11)
Cardiovascular (Cardiac disorders) | 2 (8)
Digestive (Gastrointestinal disorders) | 7 (18)
Endocrine (Endocrine disorders) | 2 (7)
General (General disorders) | 5 (8)
HEENT (Ear and labyrinth disorders) | 5 (57)
Heme & Lymphatics (Blood and lymphatic system disorders) | 11 (162)
Metabolic & Nutritional (Metabolism and nutrition disorders) | 11 (155)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 6 (15)
Nervous (Nervous system disorders) | 8 (43)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (7)
Skin & Appendages (Skin and subcutaneous tissue disorders) | 7 (12)
Urogenital (Reproductive system and breast disorders) | 4 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT00669669/Prot_SAP_000.pdf